CLINICAL TRIAL: NCT00047723
Title: Minocycline to Treat Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS045294 (NIH)
Record Dates: First submitted 2002-10-16; First posted 2002-10-17 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; amyotrophic lateral sclerosis; minocycline
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; cyclopia sequence | interventions — Minocycline

INTERVENTIONS:
Drug: minocycline

SUMMARY:
The purpose of this trial is to test the safety, tolerability, and effectiveness of minocycline compared to placebo in patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
ALS is a progressive neurodegenerative disorder without cure or known treatment that significantly improves function. Loss of motor neurons in the brain and spinal cord of ALS patients causes the progressive symptoms. Laboratory studies have linked inducible nitric oxide synthase (iNOS) and caspase enzyme activation to motor nerve cell death in ALS. Minocycline-a medication currently approved by the FDA for treatment of bacterial infections-is a tetracycline antibiotic with high central nervous system penetration when taken orally. The drug inhibits the activity of iNOS and caspase enzymes.

Minocycline has been tested and shown to protect nerve cells in many scientific experiments. It reduces cell death and prolongs survival in animal models of ALS, stroke, trauma, Huntington's disease, and Parkinson's disease. It has been shown to be beneficial in many different animal experiments of ALS, conducted in Europe, Canada and the United States.

Minocycline has been tested in 2 preliminary human trials and has been shown to be safe in patients with ALS. It has been well tolerated in conjunction with riluzole (Rilutek), the only currently FDA-approved medication for ALS.

This trial is the final important step in determining whether minocycline improves the course of ALS. The principle objective of this clinical trial is to determine whether minocycline slows disease progression and helps maintain function in patients with ALS. This multi-center placebo-controlled study will select patients early in the course of ALS, when a neuroprotective therapy may be most beneficial. The study will measure change in function (as detected by ALSFRS-R scores), strength, pulmonary function, survival, and quality of life. Participants will undergo monthly outpatient evaluations and analysis of laboratory and adverse events. This is a 13-month study.

ELIGIBILITY:
To be eligible for enrollment in this study, subjects must meet the following eligibility criteria within fourteen days prior to randomization:

Inclusion criteria:

* A clinical diagnosis of laboratory-supported probable, probable or definite ALS, according to modified EL Escorial criteria.
* FVC greater or equal to 75% of predicted.
* Onset of weakness within 3 years prior to enrollment.
* If patients are receiving riluzole they must be on a stable dose for at least the past thirty days.
* Women of childbearing age must be non-lactating and surgically sterile or using an effective method of birth control and have a negative pregnancy test (adequate birth control includes use of intra-uterine device or oral contraceptives plus a barrier method, e.g. condom, diaphragm).
* Willing and able to give signed informed consent that has been approved by your Institutional Review Board (IRB).

Exclusion criteria:

* Requirement for tracheotomy ventilation (or non-invasive ventilation > 23 hours/day).
* Diagnosis of other neurodegenerative diseases (Parkinson's disease, Alzheimer's disease, etc).
* FVC < 75% of predicted.
* A clinically significant history of unstable medical illness (unstable angina, advanced cancer, etc) over the last 30 days.
* History of renal disease (screening creatinine greater than 1.5).
* History of liver disease (screening alanine aminotransferase greater than 3 times the upper limit of normal).
* History of hematologic disease (screening white blood cell count less than 3,800/mm3).
* History of system lupus erythematosis (or screening ANA of 1:160 or greater).
* Treatment with any medications that may cause lupus-like symptoms within 4 weeks of baseline visit (e.g. procainamide, hydralazine).
* History of vestibular disease (excluding benign position vertigo).
* Pregnancy or lactation.
* Allergy to tetracycline antibiotics.
* Use of minocycline within thirty days of enrollment (baseline visit).
* Use of anti-epileptic medications other than gabapentin.
* Limited mental capacity rendering the subject unable to provide written informed consent or comply with evaluation procedures.
* History of recent alcohol or drug abuse or noncompliance with treatment or other experimental protocols.
* Use of any investigational drug within the past 30 days (Creatine, Vioxx, Celebrex, Topiramate).
* Women with the potential to become pregnant who are not practicing effective birth control.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change in function as detected by the ALS Functional Rating Scale (ALSFRS-R) in patients taking minocycline compared to those taking placebo.

SECONDARY OUTCOMES:
Changes in manual muscle testing (MMT), forced vital capacity (FVC, percent predicted), quality of life (QOL) and survival

CONTACTS AND LOCATIONS:
Overall Officials: Paul H. Gordon, M.D.,, Principal Investigator — Associate Medical Director, Eleanor and Lou Gehrig MDA/ALS Center, Columbia University Medical Center
Locations (30):
- United States (30):
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - University of California Department of Neurology, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Univ. of Colorado Health Sciences Center, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - University of Illinois, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Hennepin County Med Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - UMDNJ/Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia Unversity, Eleanor and Lou Gehrig MDA/ALS Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Metro Health Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Drexel University College of Medicine, Hahnemann Campus, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Result] Gordon PH, Moore DH, Miller RG, Florence JM, Verheijde JL, Doorish C, Hilton JF, Spitalny GM, MacArthur RB, Mitsumoto H, Neville HE, Boylan K, Mozaffar T, Belsh JM, Ravits J, Bedlack RS, Graves MC, McCluskey LF, Barohn RJ, Tandan R; Western ALS Study Group. Efficacy of minocycline in patients with amyotrophic lateral sclerosis: a phase III randomised trial. Lancet Neurol. 2007 Dec;6(12):1045-53. doi: 10.1016/S1474-4422(07)70270-3. Epub 2007 Nov 5. PMID 17980667